CLINICAL TRIAL: NCT05801952
Title: Evaluation of the Short-term Use of Selected PEP and OPEP Devices in Cystic Fibrosis Patients During an Exacerbation of the Disease
Brief Title: PEP and OPEP Devices in Cystic Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NITLD881034
Record Dates: First submitted 2023-02-15; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; PEP; OPEP
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: The 4-day physiotherapy program consists of performing bronchial drainage using one of the three devices (Aerobika* OPEP, PARI O-PEP, PARI PEP® S System). Frequency: twice a day. Physiotherapy session consist of breathing through the device for 15 breaths in one cycle, and taking a few (3-5) relaxed exhalations in accordance with the forced exhalation technique (FET). This cycle is repeated at least three times. The maximum number of cycles is five considering the need. Duration: 10 - 20 min.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobika OPEP Therapy (Experimental): Bronchial drainage session with the Aerobika OPEP device consist of breathing through the device for 15 breaths in one cycle, and taking a few (3-5) relaxed exhalations in accordance with the forced exhalation technique. This cycle is repeated at least three times. The maximum number of cycles is five considering the need. The size of the applied expiratory resistance is selected individually. The pressure is 5 - 20 cm H2O and the oscillation frequency is up to about 15 Hz. Duration of the session: 10 - 20 min. Duration of the program: 4 days. Frequency: twice a day.
  Interventions: Device: Aerobika* OPEP, PARI O-PEP (Flutter), PARI PEP® S System
- Flutter O-PEP Therapy (Experimental): Bronchial drainage session with the Flutter O-PEP device consist of breathing through the device for 15 breaths in one cycle, and taking a few (3-5) relaxed exhalations in accordance with the forced exhalation technique. This cycle is repeated at least three times. The maximum number of cycles is five considering the need. The size of the applied expiratory resistance is selected individually. The pressure is 5 - 20 cm H2O and the oscillation frequency is up to about 15 Hz. Duration of the session: 10 - 20 min. Duration of the program: 4 days. Frequency: twice a day.
  Interventions: Device: Aerobika* OPEP, PARI O-PEP (Flutter), PARI PEP® S System
- PEP Therapy (Experimental): Bronchial drainage session with the PEP device consist of breathing through the device for 15 breaths in one cycle, and taking a few (3-5) relaxed exhalations in accordance with the forced exhalation technique. This cycle is repeated at least three times. The maximum number of cycles is five considering the need. The size of the applied expiratory resistance is selected individually. The pressure is 10-20 cmH2O during exhalation. Duration of the session: 10 - 20 min. Duration of the program: 4 days. Frequency: twice a day.
  Interventions: Device: Aerobika* OPEP, PARI O-PEP (Flutter), PARI PEP® S System

INTERVENTIONS:
Device: Aerobika* OPEP, PARI O-PEP (Flutter), PARI PEP® S System — The 4-day physiotherapy program consists of performing bronchial drainage using one of the three devices: Aerobika* OPEP Device (Trudell Medical International), Flutter - PARI O-PEP Device (PARI Respiratory Equipment, Inc.) and PEP - PARI PEP® S System (PARI Respiratory Equipment, Inc.).
  Other Names: Aerobika* OPEP, Primary Device ID: 62860110504023; PARI O-PEP, Part Number: 018F65, NDC: 83490-0180-14; PARI PEP® S System, Part Number: 018F63, NDC: 83490-0180-12

SUMMARY:
Cystic fibrosis (CF) is the most common severe autosomal recessive genetic disease in Caucasians. The CFTR (cystic fibrosis transmembrane regulator) gene, which encodes the chloride channel of the epithelial cell membrane, is responsible for the development of the disease. Respiratory physiotherapy, especially bronchial drainage is one of the basic elements of comprehensive management in patients with CF. Among the many procedures used in CF drainage physiotherapy, the most commonly include these using positive expiratory pressure (PEP) and oscillating positive expiratory pressure (OPEP). The aim of the study is to assess the efficacy of the usage of selected PEP and OPEP devices in bronchial drainage in cystic fibrosis patients during exacerbation of the disease.

DETAILED DESCRIPTION:
The aim of the study is to assess the efficacy of the short-term (4-days) use of selected devices generating positive expiratory pressure (PEP device: PARI PEP® S System) and oscillating positive expiratory pressure (OPEP devices: Aerobika* OPEP Device and PARI O-PEP Device commonly called: Flutter) in bronchial drainage in cystic fibrosis patients during exacerbation of the disease. Patients will perform bronchial drainage in three different groups using different devices in each of them. The main questions study aims to answer are: 1. Whether the devices used are effective in bronchial drainage in patients with cystic fibrosis, 2. Are there differences in efficiency between the devices used.

ELIGIBILITY:
Inclusion Criteria:

* written consent of the patient and/or guardian, age over 12, no disease complications (within the last 2 months) in the form of: active haemoptysis, pneumothorax, chest surgeries, surgical procedures in the area of the esophagus (esophageal varices), otitis media,
* the ability to perform correctly lung function tests and FEV1 value above 20% predicted,
* the presence of respiratory symptoms indicating exacerbation of the disease, i.e. increasing of cough, increasing of dyspnoea, decrease in FEV1 by 10% or more from a previously recorded value.

Exclusion Criteria:

* lack of written consent of the patient and/or guardian, age below 12, occurrence of disease complications (within the last 2 months) in the form of: active hemoptysis, pneumothorax, chest surgeries, surgical procedures in the area of the esophagus (esophageal varices), otitis media,
* inability to perform lung function tests, FEV1 value below 20% of predicted value,
* PEP, OPEP device intolerance,
* no symptoms of the respiratory system indicating exacerbation of the disease, i.e. increasing of cough, increasing of dyspnoea, decrease in in FEV1 less than 10% from a previously recorded value.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function. Measured indicators: FEV1, FVC | Baseline and the day 4
  Volume measurement (L). Change from baseline to day 4
Pulmonary Function. Measured indicators: FEF75 | Baseline and the day 4
  Volume and flow measurement (L/s). Change from baseline to day 4
Sputum expectorated | from the 1st to the 4th day
  Volume measurement (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław Prusak, Principal Investigator — National Tuberculosis and Lung Diseases Research Institute
Locations (1):
- National Tuberculosis and Lung Diseases Research Institute, Rabka-Zdrój, Małopolska, Poland

REFERENCES:
- [Background] Braggion C, Cappelletti LM, Cornacchia M, Zanolla L, Mastella G. Short-term effects of three chest physiotherapy regimens in patients hospitalized for pulmonary exacerbations of cystic fibrosis: a cross-over randomized study. Pediatr Pulmonol. 1995 Jan;19(1):16-22. doi: 10.1002/ppul.1950190104. PMID 7675553
- [Result] Davies G, Rowbotham NJ, Smith S, Elliot ZC, Gathercole K, Rayner O, Leighton PA, Herbert S, Duff AJ, Chandran S, Daniels T, Nash EF, Smyth AR. Characterising burden of treatment in cystic fibrosis to identify priority areas for clinical trials. J Cyst Fibros. 2020 May;19(3):499-502. doi: 10.1016/j.jcf.2019.10.025. Epub 2019 Nov 15. PMID 31735561
- [Result] Morrison L, Innes S. Oscillating devices for airway clearance in people with cystic fibrosis. Cochrane Database Syst Rev. 2017 May 4;5(5):CD006842. doi: 10.1002/14651858.CD006842.pub4. PMID 28471492
- [Result] Lannefors L, Wollmer P. Mucus clearance with three chest physiotherapy regimes in cystic fibrosis: a comparison between postural drainage, PEP and physical exercise. Eur Respir J. 1992 Jun;5(6):748-53. PMID 1628733
- [Result] Franks LJ, Walsh JR, Hall K, Jacuinde G, Yerkovich S, Morris NR. Comparing the Performance Characteristics of Different Positive Expiratory Pressure Devices. Respir Care. 2019 Apr;64(4):434-444. doi: 10.4187/respcare.06410. Epub 2019 Jan 22. PMID 30670668
- [Result] Van Fleet H, Dunn DK, McNinch NL, Volsko TA. Evaluation of Functional Characteristics of 4 Oscillatory Positive Pressure Devices in a Simulated Cystic Fibrosis Model. Respir Care. 2017 Apr;62(4):451-458. doi: 10.4187/respcare.04570. Epub 2017 Mar 14. PMID 28292973
- [Result] Thanh NX, Jacobs P, Suggett J, McIvor A, Kaplan A. Cost-Effectiveness of the Aerobika(R) Oscillating Positive Expiratory Pressure Device in the Management of Chronic Obstructive Pulmonary Disease Exacerbations in Canada. Can Respir J. 2019 Jan 10;2019:9176504. doi: 10.1155/2019/9176504. eCollection 2019. PMID 30774739
- [Result] Leemans G, Belmans D, Van Holsbeke C, Kushnarev V, Sugget J, Ides K, Vissers D, De Backer W. A Functional Respiratory Imaging Approach to the Effect of an Oscillating Positive Expiratory Pressure Device in Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2020 Jun 4;15:1261-1268. doi: 10.2147/COPD.S242191. eCollection 2020. PMID 32581531
- [Result] Orlik T, Sands D. [Long-term evaluation of effectiveness for selected chest physiotherapy methods used in the treatment of cystic fibrosis]. Med Wieku Rozwoj. 2001 Jul-Sep;5(3):245-57. Polish. PMID 12004158
- [Result] Scherer TA, Barandun J, Martinez E, Wanner A, Rubin EM. Effect of high-frequency oral airway and chest wall oscillation and conventional chest physical therapy on expectoration in patients with stable cystic fibrosis. Chest. 1998 Apr;113(4):1019-27. doi: 10.1378/chest.113.4.1019. PMID 9554641
- [Result] Pryor JA, Webber BA, Hodson ME, Warner JO. The Flutter VRP1 as an adjunct to chest physiotherapy in cystic fibrosis. Respir Med. 1994 Oct;88(9):677-81. doi: 10.1016/s0954-6111(05)80066-6. PMID 7809441
- [Result] Chatham K, Ionescu AA, Nixon LS, Shale DJ. A short-term comparison of two methods of sputum expectoration in cystic fibrosis. Eur Respir J. 2004 Mar;23(3):435-9. doi: 10.1183/09031936.04.00084904. PMID 15065835